CLINICAL TRIAL: NCT00885820
Title: The Effects of Treatment of Subclinical Rejection on Renal Histology and Graft Function in Renal Transplant Patients Receiving Tacrolimus and Mycophenolate Mofetil
Brief Title: Benefit of Early Protocol Biopsy and Treatment of Subclinical Rejection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FKC-008
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Tacrolimus; Immunosuppression; Graft Survival
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Adrenal Cortex Hormones; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Protocol biopsies at 1, 2 and 3 months
  Interventions: Drug: Tacrolimus; Drug: MMF; Drug: Corticosteroids (Prednisone)
- 2 (Active Comparator): No protocol biopsies
  Interventions: Drug: Tacrolimus; Drug: MMF; Drug: Corticosteroids (Prednisone)

INTERVENTIONS:
Drug: Tacrolimus — Oral
  Other Names: Prograf; FK506
Drug: MMF — Oral
  Other Names: Cellcept
Drug: Corticosteroids (Prednisone) — Oral
  Other Names: Methylprednisolone; Prednisone

SUMMARY:
This multicentre randomized, controlled trial (RCT) compared renal allograft histology and function in subjects treated with Tacrolimus + MMF + prednisone undergoing early protocol biopsies and treatment of subclinical rejection versus a non-protocol biopsy control group.

ELIGIBILITY:
Inclusion Criteria:

* Subject is the recipient of a first or second cadaveric or living donor mismatched (at least one mismatch) renal transplant
* If female and of child-bearing potential, subject has a negative pregnancy test and utilizes adequate contraceptive methods

Exclusion Criteria:

* Recipients of a kidney from a donor over 65 years of age
* Recipient of non-related donor kidney with peak pre-transplant PRA > 50
* Subject has lost a previous graft to rejection less than one year from transplant
* Subject who has received an investigational drug within three months prior to randomization
* Subjects who are pregnant or breastfeeding
* Subject receives a kidney lacking a pre-implantation biopsy
* Subject has significant disease or disability (e.g. malignancy or uncontrolled infection) which prevents adherence to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2001-09; Primary Completion 2004-07 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The incidence of interstitial fibrosis/tubular atrophy as defined by Banff interstitial and tubular chronic changes of ci + ct of 2 or more at 6 months | 6 months

SECONDARY OUTCOMES:
The incidence of subclinical rejection at 6 months | 6 months
Prevalence of chronic renal histopathology at 24 months | 24 months
Renal function as determined by serum creatinine and 24 hour urine creatinine clearance and protein excretion | 6, 12 and 24 moths

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Canada, Inc.
Locations (10):
- Palo Alto, California, United States
- Canada (9):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Background] Rush DN, Cockfield SM, Nickerson PW, Arlen DJ, Boucher A, Busque S, Girardin CE, Knoll GA, Lachance JG, Landsberg DN, Shapiro RJ, Shoker A, Yilmaz S. Factors associated with progression of interstitial fibrosis in renal transplant patients receiving tacrolimus and mycophenolate mofetil. Transplantation. 2009 Oct 15;88(7):897-903. doi: 10.1097/TP.0b013e3181b723f4. PMID 19935461